CLINICAL TRIAL: NCT04671576
Title: Evaluation of Growth and Safety of Healthy Term Infants Consuming an Organic Formula.
Brief Title: Growth and Safety Clinical Trial on a New Infant Formula.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nara Organics (Industry)
Collaborators: Paidion Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NA-101-19
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: Healthy Growth
Keywords: infant formula; cow milk; growth

STUDY DESIGN:
Intervention Model Description: A controlled, decentralized, double-blind trial of healthy, term, formula-fed infants randomized to one of two infant formulas:
  Control Formula (a standard, commercially available infant formula) or Investigational Formula for 16 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Formula (Active Comparator): A standard, milk-based, infant formula.
  Interventions: Other: Control Infant Formula
- Investigational Formula (Experimental): An organic milk-based infant formula.
  Interventions: Other: Organic Infant Formula

INTERVENTIONS:
Other: Control Infant Formula — Powder, standard commercial infant formula.
  Arms: Control Formula
Other: Organic Infant Formula — Powder, organic milk-based infant formula.
  Arms: Investigational Formula

SUMMARY:
The aim of the study is to assess age-appropriate growth of healthy infants fed a new organic milk-based infant formula.

DETAILED DESCRIPTION:
A 16-weeks length, randomized, controlled, double-blind, parallel study designed to evaluate growth and tolerance of healthy infants fed milk-based infant formula. The study has been designed in accordance with Good Clinical Practice guidelines and the requirements of the Code of Federal Regulations 21 CFR 106.96

ELIGIBILITY:
Inclusion Criteria:

* Healthy gestational term (≥ 37 wks; ≤ 41 wks and 6 days).
* Birth weight of ≥ 2,500 g and ≤ 4,500 g.
* Postnatal age ≤ 14 days.
* Singleton.
* Designated as healthy, that is no recognized diseases.
* Weight, length, weight-for-length, and head circumference within ≥ 5th and ≤ 95th percentile for age-sex according to World Health Organization (WHO) growth standards (birth to 24 months).
* Exclusive feeding and tolerating cow milk formula at time of enrollment.
* Parent(s) or legal guardians are willing and able to feed the assigned formula as sole source of nutrition.
* Parent(s) or legal guardians are willing and able to participate in anthropometric procedures.
* Parent(s) or legal guardians have voluntarily signed and dated required participation forms, such as the ICF approved by an IRB.

Exclusion Criteria:

* An infant from a multiple birth, such as twin, triplet, or the like.
* Personal or immediate family history of cow-milk protein allergy or intolerance.
* Currently on any medication to treat growth failure or that may significantly impact growth.
* Evidence of any anatomic and/or physiologic condition that would interfere with normal growth, development, or feeding, such as genetic, neurological, gastrointestinal, cardiac, pulmonary, hepatic, or renal.
* A maternal history with known adverse effects on the fetus and/or the newborn infant, such as positive HIV, insulin-dependent diabetes, opioid exposure during pregnancy.
* Enrolled in another clinical trial involving a drug, nutrition supplement, device, or intervention.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Formula intake. | Study Day 1 to Study Day 112
  Volume of formula consumed. ml/day
Weight. | Study Day 1 to Study Day 112
  Weight. Weight gain velocity. g and g/day
Length. | Study Day 1 to Study Day 112
  Length. Length gain velocity. cm and cm/day.
Head circumference. | Study Day 1 to Study Day 112
  Head circumference. Head circumference gain velocity. cm and cm/day
Anthropometry Z-scores. | Study Day 1 to Study Day 112
  Weight for age Z-score. Length for age Z-score. Weight for length Z-score. Head circumference for age Z-score.

SECONDARY OUTCOMES:
Formula tolerance. | Study Day 1 to Study Day 112
  Frequency of adverse events. Fussiness. Inconsolable crying.
Gastrointestinal characteristic. | Study Day 1 to Study Day 112
  Stool consistency. Stools/day. Regurgitation. Gas.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Fingarson, DO, Study Director — Paidion Research, Inc.; Tiffany Petty, MD, Principal Investigator — Telehub Research
Locations (1):
- TeleResearch Hub, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No